CLINICAL TRIAL: NCT01215591
Title: Randomized Controlled Trial of Gradual Versus Sudden Weaning From Nasal CPAP in Preterm Neonates
Brief Title: Trial of Weaning of Nasal Continuous Positive Airway Pressure (CPAP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, Shantanu Rastogi, Neonatologist, Maimonides Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Maimonides Project 07/10/VA5
Record Dates: First submitted 2010-09-27; First posted 2010-10-06 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Preterm Neonates
Keywords: Neonatal; Nasal CPAP; Randomized controlled trial; Weaning
MeSH Terms: interventions — Weaning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gradual wean from Nasal CPAP (Active Comparator): Nasal CPAP for gradual wean group it was cycled off for 3 hours alternating with 3 hours on for first 48 hours, if successful the cycle was extended to 6 hours off and 3 hours on for the next 48 hours. If the baby tolerated this regime the prongs were removed and CPAP was kept off.
  Interventions: Procedure: Gradual weaning from Nasal CPAP in preterm neonates
- Sudden wean from Nasal CPAP (No Intervention): Usual practice to wean the preterm neonates from nasal CPAP

INTERVENTIONS:
Procedure: Gradual weaning from Nasal CPAP in preterm neonates — Nasal CPAP for gradual wean group it was cycled off for 3 hours alternating with 3 hours on for first 48 hours, if successful the cycle was extended to 6 hours off and 3 hours on for the next 48 hours. If the baby tolerated this regime the prongs were removed and CPAP was kept off.
  Other Names: Nasal CPAP; Weaning; Preterm neonates
  Arms: Gradual wean from Nasal CPAP

SUMMARY:
To compare the 2 methods of weaning of nasal CPAP in premature babies born at 32 weeks or less

DETAILED DESCRIPTION:
Objective: To study the weight and the post menstrual age (PMA) at the time of nasal CPAP (NCPAP) wean utilizing the method of sudden wean as compared to gradual wean. . Methods: A prospective randomized trial was conducted comparing sudden weaning with gradual weaning from NCPAP in neonates with gestational age (GA) <32 weeks. The patients were randomized to one of the two methods of weaning from NCPAP and their success was compared.

ELIGIBILITY:
Inclusion Criteria:

All babies born with GA <32 weeks admitted to the neonatal intensive care units at the Maimonides Infant and Children's Hospital, between 1st January 2008 and 31st March 2009 and required to be on NCPAP for longer than 48 hours.-

Exclusion Criteria:

Those with severe congenital anomalies and chromosomal defects including congenital heart disease and neurological malformations, chest wall or airway abnormalities and lung hypoplasia, were excluded from the cohort

Ages: 24 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Weight when preterm neonates could come off nasal CPAP | During the initial NICU stay
  Weight when preterm neonates could come off nasal CPAP
Post-menstrual age when preterm neonates could come off nasal CPAP | During the initial NICU stay
  Post-menstrual age when preterm neonates could come off nasal CPAP

SECONDARY OUTCOMES:
Weights when the neonates could come off oxygen | During the initial NICU stay
  Weights when the neonates could come off oxygen
length of stay in the hospital | During the initial NICU stay
  length of stay in the hospital
Post-menstrual age when preterm neonates could come off oxygen | During the initial NICU stay
  Post-menstrual age when preterm neonates could come off oxygen

CONTACTS AND LOCATIONS:
Overall Officials: Shantanu Rastogi, MD, Principal Investigator — Maimonides Medical Center; Alok Bhutada, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

REFERENCES:
- See also: pubmed abstract — http://www.ncbi.nlm.nih.gov/pubmed/22906960